CLINICAL TRIAL: NCT01211262
Title: A Phase 1, Open Label, Dose Finding Study to Assess the Safety and Tolerability of IMCgp100, a Monoclonal T Cell Receptor Anti-CD3 scFv Fusion Protein in Patients With Advanced Malignant Melanoma
Brief Title: Study to Assess the Tolerability of a Bispecific Targeted Biologic IMCgp100 in Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100/01; 2010-019290-15 (EudraCT Number)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Phase I; Biologic
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMCgp100 weekly dosing regimen (Experimental): Weekly intravenous (IV) infusions of IMCgp100 over treatment cycles of 8 weeks each.
  Interventions: Drug: IMCgp100
- IMCgp100 daily dosing regimen (Experimental): Daily IV infusions of IMCgp100 administered on days 1 to 4 and days 22 to 25 of a six-week treatment cycle.
  Interventions: Drug: IMCgp100

INTERVENTIONS:
Drug: IMCgp100 — For each arm, the study will be divided into two parts: In part 1, dose escalation, the MTD or RP2D for each dosing regimen will be established. In part 2, dose expansion, a cohort of participants will be treated at the RP2D or MTD.
  Other Names: ImmTACgp100

SUMMARY:
IMCgp100 is a new biological therapy designed for the treatment of melanoma skin cancer. The drug is designed to target melanoma cells and stimulate immune cells to kill them. This trial is designed to establish the level of drug that can be given to a patient that is tolerable. It also designed to establish the best dosing schedule for the drug and to look for signals that the drug is working as intended.

DETAILED DESCRIPTION:
IMCgp100 is a bispecific biologic incorporating an engineered T cell receptor (TCR) specific for a peptide antigen derived from the protein gp100 presented in the context of HLA A2 on the surface of melanoma cells. The TCR is fused to an anti-CD3 antibody single-chain variable fragment (scFv) that recruits and activates non-melanoma specific T cells (killer T cells) in physical contact with the cancer T cell. This is a Phase I study designed to assess the safety profile and establish a tolerable dose of IMCgp100 in HLA A2 positive malignant melanoma patients. The study has two treatment arms with different treatment schedules, weekly or daily dosing. Each treatment arm in the study has two parts. In the first part, dose escalation, the safety and tolerability of the drug are examined and the optimal dose of drug is established. In the second part of the trial, participants will receive an extended course of treatment with a view to assessing the effect of the drug on disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically documented Stage IV malignant melanoma or unresectable Stage III melanoma for which no standard effective therapy exists or for which an appropriate window exists between alternative therapeutic options. Participants for whom early treatment with vemurafenib is indicated, e.g. rapidly progressing or symptomatic disease, are excluded from this trial.
2. Previous surgery (other than resection of skin metastases), radiotherapy, chemotherapy, immunotherapy or experimental therapy completed > 4 weeks before and all adverse events resolved to ≤ grade 1. In cases where localized radiotherapy has been applied, treatment with IMCgp100 can be commenced after a two week period.
3. Human leukocyte antigen (HLA) A2 positive.
4. ≥ 18 years old.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. Participants participating in the dose escalation part of Arm 2 only require assessable disease.
7. Life expectancy > 3 months.
8. Blood tests within the following parameters:

   1. Platelet count ≥ 100 x10⁹/L
   2. Hemoglobin ≥ 9g/dL (blood transfusion to achieve this level is permitted)
   3. Calculated creatinine clearance ≥ 50 mL/min using the modified Cockroft-Gault equation
   4. Neutrophil count ≥1x10⁹/L
   5. Lymphocyte count ≥ 0.5x10⁹/L
9. Female participants of childbearing potential must use maximally effective birth control during the period of therapy, must be willing to use contraception for 6 months following the last study drug infusion and must have a negative urine or serum pregnancy test upon entry into this study. Otherwise, female participants must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile.
10. Male participants must be surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 6 months following the last study drug infusion.
11. Participants with a history of adrenal insufficiency, maintained on stable replacement dose corticosteroid (< 10 mg/d prednisone or the equivalent) are eligible for treatment with IMCgp100, unless there is a past history of adrenal crisis. Eligible participants with a history of adrenal insufficiency receiving replacement dose corticosteroid must receive prophylactic stress dose corticosteroid prior to dosing during the first four doses of IMCgp100 treatment, regardless of weekly or daily dosing regimen.
12. Able to give informed consent.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Symptomatic brain metastases that are unstable, require steroids, or that have required radiation within the last 28 days.
2. Other active malignancy in the past 5 years except carcinoma in situ, completely excised nonmelanomatous skin cancer or any other malignancy that in the opinion of the investigator is considered to be cured.
3. Comorbid medical condition that would increase the risk of toxicity in the opinion of the investigator or sponsor. Symptomatic on-going infection must be resolved before the patient can be treated in the study.
4. Uveitis.
5. Had myocardial infarction within 1 year before enrolment, symptomatic congestive heart failure (New York Heart Association > Class II), unstable angina or unstable cardiac arrhythmia requiring medication.
6. Has an ejection fraction < 50%.
7. Clinically significant electrocardiogram (ECG) changes that obscure the ability to assess the RR, PR and QT intervals. Participants with corrected QT interval (QTc) calculated by Bazetts or locally preferred formula which is greater than 500 ms.
8. Has hepatic function as follows:

   1. Aspartate aminotransferase > 2.5 x upper limit of normal (ULN)
   2. Alanine aminotransferase > 2.5 x ULN
   3. Bilirubin > 2.0 x ULN
   4. Prothrombin time or partial thromboplastin time > 1.5 x ULN
9. Bleeding diathesis
10. Immunosuppressive condition or treatment including previous transplantation, splenectomy or known human immunodeficiency virus (HIV) infection.
11. Has a history of adult seizures.
12. Participants with evidence of a raised intracranial pressure in Arm 2 of the study who will have a cerebrospinal fluid sample taken.
13. Participants receiving chronic corticosteroid treatment (longer than 8 weeks duration) for management of pre-existing adverse events at any dose, or participants with a history of chronic corticosteroid treatment longer than 8 weeks duration for adverse events within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namir Hassan, PhD, Study Director — Immunocore Ltd
Locations (9):
- United States (4):
  - The Angeles Clinic, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Slone Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - The Beatson Institute, Glasgow
  - St James Hospital, Leeds
  - NIHR Biomedical Research Centre, Oxford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All-patients population and safety population both comprised 84 participants who enrolled in the study and who also received at least one IMCgp100 dose; the all-patients and safety population for Arm 1 was 66 participants and for Arm 2 was 18 participants. Efficacy population was 54 participants in Arm 1 and 15 participants in Arm 2.
Period: Overall Study
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Started | 66 | 18
Completed | 43 | 8
Not Completed | 23 | 10
Not completed — Progressive Disease | 18 | 9
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: The all-patients population and the safety population both comprised the 84 participants who enrolled in the study and who also received at least one IMCgp100 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen | Total
Number analyzed (Participants) | 66 | 18 | 84
Age, Continuous [Mean (Full Range); unit: years] | 58.2 [25 to 78] | 60.4 [31 to 75] | 58.7 [25 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 5 | 30
  Male | 41 | 13 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62 | 17 | 79
  Black | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of IMCgp100 Administered Weekly (Dose Escalation Part)
Description: The maximum tolerated dose (MTD) for IMCgp100 administered by weekly dosing was determined based on the frequency of dose-limiting toxicity (DLT) occurring during Days 1 to 8. Participants presented at MTD in the dose escalation phase.
  Abbreviations: ng/kg=nanograms/kilogram
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
Population: Safety population: all participants who received at least 1 dose of IMCgp100, up to a maximum of 600 ng/kg.
Measure: Number; unit: ng/kg
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 27
ng/kg | 600

2. Primary Outcome: MTD of IMCgp100 Administered Daily (Dose Escalation Part)
Description: The MTD for IMCgp100 administered by daily dosing was determined based on the frequency of DLT occurring during Days 1 to 8. The 50 mcg dose was the RP2D for daily dosing, as the MTD was not achieved.
  Abbreviations: mcg=micrograms
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
Population: Safety population: all participants who received at least 1 dose of IMCgp100
Measure: Number; unit: mcg
Groups:
- IMCgp100 Daily Dosing Regimen: Daily intravenous (IV) infusions of IMCgp100 over treatment cycles of 8 weeks each.
Arm/Group | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 18
mcg | 50

3. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) with an onset date after the date of first dose and within 30 days after the last administration of study medication in either treatment arm. AEs with missing date of onset were considered treatment emergent.
Time Frame: Day 1 (first dose), 30 days after the last dose
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
percentage of participants | 100.0 | 100.00

4. Primary Outcome: Number of Participants Experiencing Clinically Significant Laboratory Parameters (Hematology)
Description: Laboratory parameters included clinical chemistry, hematology, and urinalysis. For hematology, this included red cell count, hemoglobin, hematocrit, mean cell volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, leukocyte differential count (percentage or absolute), prothrombin time, and activated partial tissue thromboplastin time. Clinically significant findings were defined as such in the opinion of the investigator occurring at any time on treatment from normal pre-dose.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Groups:
- IMCgp100 Daily Dosing Regimen: Daily IV infusions of IMCgp100 administered on days 1 to 4 and days 22 to 25 of a six-week treatment.
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants
  Lymphocytes | 12 | 1
  Hemoglobin | 1 | 2
  Neutrophils | 1 | 0
  CD4 Cells | 1 | 0
  Leukocytes | 1 | 0

5. Primary Outcome: Number of Participants Experiencing ≥Grade 3 Severity in Laboratory Parameters (Hematology)
Description: Laboratory parameters included clinical chemistry, hematology, and urinalysis. For hematology, this included red cell count, hemoglobin, hematocrit, mean cell volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, leukocyte differential count (percentage or absolute), prothrombin time, and activated partial tissue thromboplastin time. Laboratory parameter abnormalities were graded by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 at any time on treatment from normal pre-dose. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants
  Lymphocytes-Grade 3: number analyzed (Participants) | 61 | 16
  Lymphocytes-Grade 3 | 15 | 2
  Lymphocytes-Grade 4: number analyzed (Participants) | 61 | 16
  Lymphocytes-Grade 4 | 2 | 2
  CD4 Count-Grade 3: number analyzed (Participants) | 32 | 1
  CD4 Count-Grade 3 | 4 | 1
  CD4 Count-Grade 4: number analyzed (Participants) | 32 | 1
  CD4 Count-Grade 4 | 4 | 1
  Hemoglobin-Grade 3: number analyzed (Participants) | 63 | 17
  Hemoglobin-Grade 3 | 0 | 3
  Leukocytes-Grade 3: number analyzed (Participants) | 65 | 17
  Leukocytes-Grade 3 | 1 | 0

6. Primary Outcome: Number of Participants Experiencing Clinically Significant Laboratory Parameters (Clinical Chemistry)
Description: Laboratory parameters included clinical chemistry, hematology, and urinalysis. Clinical chemistry parameters included calcium, phosphorus, magnesium, albumin, bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, lactate dehydrogenase, sodium, potassium, bicarbonate, creatinine, chloride, glucose, urea, uric acid, and C-reactive protein. Clinically significant findings were defined as such in the opinion of the investigator occurring at any time on treatment from normal pre-dose.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants
  Albumin | 3 | 3
  Alkaline Phosphatase | 3 | 1
  Aspartate Aminotransferase | 1 | 2
  Alanine Aminotransferase | 1 | 1
  Potassium | 1 | 1
  Calcium | 0 | 1
  Glucose | 1 | 0
  Magnesium | 0 | 1
  Sodium | 0 | 1
  Uric Acid | 1 | 0

7. Primary Outcome: Number of Participants Experiencing ≥Grade 3 Severity in Laboratory Parameters (Clinical Chemistry)
Description: Laboratory parameters included clinical chemistry, hematology, and urinalysis. Clinical chemistry parameters included calcium, phosphorus, magnesium, albumin, bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, lactate dehydrogenase, sodium, potassium, bicarbonate, creatinine, chloride, glucose, urea, uric acid, and C-reactive protein. Laboratory parameter abnormalities were graded by the investigator using CTCAE v 4.0 at any time on treatment from normal pre-dose. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants
  Sodium-Grade 3: number analyzed (Participants) | 62 | 18
  Sodium-Grade 3 | 2 | 4
  Potassium-Grade 3: number analyzed (Participants) | 62 | 17
  Potassium-Grade 3 | 2 | 1
  Glucose-Grade 3: number analyzed (Participants) | 63 | 17
  Glucose-Grade 3 | 1 | 1
  Aspartate Aminotransferase-Grade 3: number analyzed (Participants) | 63 | 18
  Aspartate Aminotransferase-Grade 3 | 1 | 0
  Calcium-Grade 3: number analyzed (Participants) | 64 | 18
  Calcium-Grade 3 | 0 | 1

8. Primary Outcome: Number of Participants Experiencing Clinically Significant Electrocardiograms (ECGs)
Description: Twelve lead ECGs were obtained after the participant has rested in a supine position for at least 5 minutes. Clinically significant findings were defined as such in the opinion of the investigator or designated physician occurring at any time on treatment from normal pre-dose.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants | 3 | 0

9. Primary Outcome: Number of Participants Experiencing Clinically Significant Vital Signs
Description: Vital signs included temperature, blood pressure, respiration rate, and heart rate. Measurements were made after the participant had been resting supine for a minimum of 5 minutes. Blood pressure and heart rate were measured using a recording device with an appropriate cuff size. Temperature and respiration rate were measured as per clinical practice. Clinically significant findings were defined as such in the opinion of the investigator occurring at any time on treatment from normal pre-dose.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants
  High Systolic Blood Pressure | 17 | 2
  Low Systolic Blood Pressure | 8 | 5
  High Diastolic Blood Pressure | 20 | 3
  Low Diastolic Blood Pressure | 37 | 12
  High Heart Rate | 34 | 12
  Low Heart Rate | 8 | 1
  High Temperature | 33 | 13

10. Primary Outcome: Number of Participants Experiencing Clinically Significant Physical Examination Results (Weight Decrease)
Description: Physical examination included weight, a record of skin pigmentation, and photographic record of any vitiligo if present. Clinically significant findings were defined as such in the opinion of the investigator occurring at any time on treatment from normal pre-dose.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants | 3 | 1

11. Primary Outcome: Number of Participants Experiencing ≥Grade 3 Severity in Physical Examination Results (Skin Pigmentation)
Description: Physical examination included weight, a record of skin pigmentation, and photographic record of any vitiligo if present. Abnormalities were graded by the investigator using CTCAE v 4.0 at any time on treatment from normal pre-dose. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death.
Time Frame: 28 months
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
number of participants | 0 | 0

12. Secondary Outcome: Number of Participants With Best Overall Response Per Response Evaluation Criteria In Solid Tumors (RECIST) (Weekly Dosing-Dose Expansion Part)
Description: The best overall response was assigned as complete response (CR), partial response (PR), minor response, stable disease, progressive disease (PD) or not evaluable (NE) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Time Frame: 28 months
Population: Efficacy population: only evaluable participants (those having both a baseline and post treatment sample).
Measure: Number; unit: participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 54 | 15
participants | 5 | 1

13. Secondary Outcome: Number of Participants With Anti-IMCgp100 Antibody Formation (Dose Escalation and Dose Expansion Parts)
Description: To provide a comprehensive anti-drug antibody (ADA) summary for the study, individual participant data were combined and assessed as distinct groups based on characteristics of their ADA response. Evaluable participants were those with post-drug administration samples. ADA prevalence (pre- existing antibody response) was measured as the number of baseline-positive participant out of all participants who provided baseline samples. Overall ADA incidence was calculated based on the combined number of treatment-boosted and treatment-induced ADA-positive participants. The treatment-induced incidence was determined as the number of ADA- positive participants of those that were ADA-negative at baseline; while treatment-boosted incidence was determined as the number of participants with an ADA titer increase equal to or greater than the minimum significant dilution (3-fold) of the assay.
Time Frame: 28 months
Population: Efficacy population
Measure: Number; unit: participants
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 66 | 18
participants | 2 | 1

14. Secondary Outcome: Estimated Maximum Plasma Concentration (Cmax) of IMCgp100 By-weight Doses (Dose Escalation)
Description: The maximum plasma concentration (Cmax) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. Abbreviations: ng/kg = nanograms/kilogram
Time Frame: Day 1, Cycle 1
Population: Pharmacokinetics (PK) Population: all participants who receive at least 1 dose of IMCgp100 and have at least 1 measurable PK concentration with the relevant date, time and dosing data for this sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 42
picograms/milliliter
  15 ng/kg by-weight dose: number analyzed (Participants) | 3
  15 ng/kg by-weight dose | 305.50 (583.47)
  45 ng/kg by-weight dose: number analyzed (Participants) | 3
  45 ng/kg by-weight dose | 271.33 (21.49)
  135 ng/kg by-weight dose: number analyzed (Participants) | 3
  135 ng/kg by-weight dose | 371.79 (57.25)
  270 ng/kg by-weight dose: number analyzed (Participants) | 3
  270 ng/kg by-weight dose | 856.35 (41.01)
  405 ng/kg by-weight dose: number analyzed (Participants) | 6
  405 ng/kg by-weight dose | 2345.25 (35.74)
  600 ng/kg by-weight dose: number analyzed (Participants) | 20
  600 ng/kg by-weight dose | 6188.54 (41.21)
  900 ng/kg by-weight dose: number analyzed (Participants) | 4
  900 ng/kg by-weight dose | 8868.83 (27.92)

15. Secondary Outcome: Estimated Cmax of IMCgp100 of 900 ng/kg By-weight Dose (Dose Escalation and Dose Expansion Parts)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 4
picograms/milliliter | 8868.83 (27.92)

16. Secondary Outcome: Estimated Cmax of IMCgp100 Flat Dose (Dose Escalation and Dose Expansion Parts)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval. Abbreviations: mcg = micrograms
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 21
picograms/milliliter
  20 mcg: number analyzed (Participants) | 7
  20 mcg | 3239.82 (20.97)
  40 mcg: number analyzed (Participants) | 3
  40 mcg | 8316.43 (45.10)
  50 mcg: number analyzed (Participants) | 11
  50 mcg | 8740.99 (38.01)

17. Secondary Outcome: Estimated Cmax of IMCgp100 of 600 ng/kg By-weight Dose (Dose Escalation)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Cycle 1: Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50
Population: PK Population
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 10
picograms/milliliter
  Day 1 | 7311 (1770)
  Day 8: number analyzed (Participants) | 9
  Day 8 | 5726 (3605)
  Day 15: number analyzed (Participants) | 9
  Day 15 | 6182 (1456)
  Day 22: number analyzed (Participants) | 9
  Day 22 | 6490 (2488)
  Day 29: number analyzed (Participants) | 9
  Day 29 | 6245 (3047)
  Day 36: number analyzed (Participants) | 9
  Day 36 | 6396 (3474)
  Day 43: number analyzed (Participants) | 8
  Day 43 | 6014 (1125)
  Day 50: number analyzed (Participants) | 8
  Day 50 | 7136 (2744)

18. Secondary Outcome: Estimated Cmax of IMCgp100 of 20/30/50 mcg Flat Dose (Dose Escalation)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval. On Day 1, IMCgp100 20 mcg was given, IMCgp100 30 mcg was administered on Day 8, and IMCgp100 50 mcg was dosed on Days 15 and after.
Time Frame: Cycle 1: Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50
Population: PK Population
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 7
mcg
  Day 1 | 3299 (660)
  Day 8 | 5056 (1175)
  Day 15 | 7981 (2278)
  Day 22: number analyzed (Participants) | 6
  Day 22 | 6682 (1395)
  Day 29 | 4710 (3621)
  Day 36: number analyzed (Participants) | 5
  Day 36 | 7100 (1535)
  Day 43 | 7240 (1906)
  Day 50: number analyzed (Participants) | 6
  Day 50 | 6658 (1211)

19. Secondary Outcome: Estimated Cmax of IMCgp100 of 40/40/50 mcg Flat Dose (Dose Escalation)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval. This dosing regimen was implemented following the Urgent Safety Measure to adapt the dosing in the Phase 1 study that dropped Dose 1 to 40 mcg from the identified 50 mcg RP2D.
Time Frame: Cycle 1: Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50
Population: PK Population
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 3
mcg
  Day 1 | 8847 (3811)
  Day 8: number analyzed (Participants) | 2
  Day 8 | 5340 (311)
  Day 15 | 8373 (2682)
  Day 22: number analyzed (Participants) | 2
  Day 22 | 7445 (983)
  Day 29: number analyzed (Participants) | 2
  Day 29 | 3288 (4614)
  Day 36 | 8073 (1337)
  Day 43: number analyzed (Participants) | 2
  Day 43 | 6735 (672)
  Day 50: number analyzed (Participants) | 2
  Day 50 | 7130 (4483)

20. Secondary Outcome: Estimated Cmax of IMCgp100 of 50 mcg Flat Dose (Dose Escalation)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The RP2D identified in this study following review of all safety and pharmacokinetic data in the dose escalation of the Phase 1 study was the 50 mcg flat dose.
Time Frame: Cycle 1: Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50
Population: PK Population
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 11
mcg
  Day 1 | 9327 (3802)
  Day 8: number analyzed (Participants) | 8
  Day 8 | 6414 (3653)
  Day 15: number analyzed (Participants) | 10
  Day 15 | 7236 (3304)
  Day 22: number analyzed (Participants) | 10
  Day 22 | 7620 (2710)
  Day 29: number analyzed (Participants) | 9
  Day 29 | 8186 (3178)
  Day 36: number analyzed (Participants) | 10
  Day 36 | 8425 (4594)
  Day 43: number analyzed (Participants) | 9
  Day 43 | 6905 (4097)
  Day 50: number analyzed (Participants) | 9
  Day 50 | 9018 (5001)

21. Secondary Outcome: Estimated Cmax of IMCgp100 of a Single Infusion Flat Dose (Dose Escalation)
Description: The Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Cycle 1: Day 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter
Arm/Group | IMCgp100 Daily Dosing Regimen
Number analyzed (Participants) | 18
picograms/milliliter
  10 mcg: number analyzed (Participants) | 3
  10 mcg | 997.83 (38.01)
  20 mcg: number analyzed (Participants) | 3
  20 mcg | 3599.18 (15.42)
  30 mcg: number analyzed (Participants) | 3
  30 mcg | 3599.18 (15.42)
  40 mcg: number analyzed (Participants) | 4
  40 mcg | 6157.90 (29.52)
  50 mcg: number analyzed (Participants) | 5
  50 mcg | 8111.79 (27.80)

22. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of IMCgp100 By-weight Dose (Dose Escalation)
Description: The area under the concentration-time curve (AUC), measured in hours by picograms per milliliter ( h*pg/ml) is a method of measurement of the total exposure of a drug in blood.
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 42
hours * picograms/milliliter
  15 ng/kg: number analyzed (Participants) | 3
  15 ng/kg | 5666.63 (434.62)
  45 ng/kg: number analyzed (Participants) | 3
  45 ng/kg | 2965.10 (49.17)
  135 ng/kg: number analyzed (Participants) | 3
  135 ng/kg | 2904.91 (96.95)
  270 ng/kg: number analyzed (Participants) | 3
  270 ng/kg | 10649.19 (40.82)
  405 ng/kg: number analyzed (Participants) | 6
  405 ng/kg | 33332.31 (43.57)
  600 ng/kg: number analyzed (Participants) | 20
  600 ng/kg | 63507.24 (43.97)
  900 ng/kg: number analyzed (Participants) | 4
  900 ng/kg | 97724.58 (29.49)

23. Secondary Outcome: AUC of IMCgp100 of 900 ng/kg By-weight Dose (Dose Escalation and Dose Expansion Parts)
Description: The AUC, measured in h*pg/ml, is a method of measurement of the total exposure of a drug in blood.
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 4
hours * picograms/milliliter | 97724.58 (29.49)

24. Secondary Outcome: AUC of IMCgp100 Flat Dose (Dose Escalation and Dose Expansion Parts)
Description: The AUC (measured in h*pg/ml) is a method of measurement of the total exposure of a drug in blood. Participants in the 20 mcg and 40 mcg dose groups received intra-participant dose-escalation up to 50 mcg on Day 15.
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 10
hours * picograms/milliliter
  20 mcg: number analyzed (Participants) | 7
  20 mcg | 3239.82 (20.97)
  40 mcg: number analyzed (Participants) | 3
  40 mcg | 59333.15 (21.44)

25. Secondary Outcome: AUC of IMCgp100 of 50 mcg Flat Dose (Dose Escalation and Dose Expansion Parts)
Description: The AUC (measured in h*pg/ml) is a method of measurement of the total exposure of a drug in blood.
Time Frame: Day 1, Cycle 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * picograms/milliliter
Arm/Group | IMCgp100 Weekly Dosing Regimen
Number analyzed (Participants) | 11
hours * picograms/milliliter | 73134.57 (55.88)

ADVERSE EVENTS:
Time Frame: Up to Day 80 (follow up)
Description: Adverse events were recorded from the time informed consent was obtained to 30 days after the final dose or 30 days after withdrawal from treatment. The safety population was comprised of the 84 participants who enrolled in the study and included all participants who received at least one dose of IMCgp100.
Groups:
- IMCgp100 Weekly Dosing Regimen: Weekly intravenous (IV) infusions of IMCgp100 at the weekly maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) over treatment cycles of eight weeks each.
- IMCgp100 Daily Dosing Regimen: Daily IV infusions of IMCgp100 administered on days 1 to 4 and days 22 to 25 of a six week treatment cycle at the MTD/daily RP2D.
Arm/Group | IMCgp100 Weekly Dosing Regimen | IMCgp100 Daily Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 8/66 | 8/18
Serious Adverse Events (participants affected / at risk) | 24/66 | 5/18
Other Adverse Events (participants affected / at risk) | 66/66 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMCgp100 Weekly Dosing Regimen (N=66) | IMCgp100 Daily Dosing Regimen (N=18)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 2 (2) | 0 (0)
DISEASE PROGRESSION (General disorders) | 2 (2) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1 (1) | 0 (0)
BILIARY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTRIC INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LABORATORY TEST ABNORMAL (Investigations) | 1 (1) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 2 (3) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 4 (5) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMCgp100 Weekly Dosing Regimen (N=66) | IMCgp100 Daily Dosing Regimen (N=18)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 13 (13) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
SINUS TACHYCARDIA (Cardiac disorders) | 5 (5) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 7 (7) | 4 (4)
ERYTHEMA OF EYELID (Eye disorders) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 0 (0) | 1 (1)
EYE PAIN (Eye disorders) | 2 (2) | 1 (1)
EYELID OEDEMA (Eye disorders) | 0 (0) | 1 (1)
OCULAR HYPERAEMIA (Eye disorders) | 2 (2) | 1 (1)
PERIORBITAL OEDEMA (Eye disorders) | 30 (30) | 11 (11)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (9) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 14 (14) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 10 (10) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 34 (34) | 10 (10)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 24 (24) | 10 (10)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
AXILLARY PAIN (General disorders) | 2 (2) | 1 (1)
CHEST PAIN (General disorders) | 7 (7) | 0 (0)
CHILLS (General disorders) | 17 (17) | 9 (9)
FACE OEDEMA (General disorders) | 13 (13) | 3 (3)
FATIGUE (General disorders) | 35 (35) | 10 (10)
INFLUENZA LIKE ILLNESS (General disorders) | 13 (13) | 5 (5)
MALAISE (General disorders) | 2 (2) | 1 (1)
OEDEMA (General disorders) | 4 (4) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 10 (10) | 8 (8)
PAIN (General disorders) | 2 (2) | 2 (2)
PERIPHERAL SWELLING (General disorders) | 6 (6) | 2 (2)
PYREXIA (General disorders) | 34 (34) | 13 (13)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1)
ANGULAR CHEILITIS (Infections and infestations) | 4 (4) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 5 (5) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1)
RHINITIS (Infections and infestations) | 6 (6) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (3) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 3 (3)
WEIGHT DECREASED (Investigations) | 1 (1) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 (9) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 (14) | 2 (2)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4) | 0 (0)
HEADACHE (Nervous system disorders) | 16 (16) | 6 (6)
LETHARGY (Nervous system disorders) | 5 (5) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 10 (10) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RALES (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 18 (18) | 5 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 17 (17) | 2 (2)
GENERALISED ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 43 (43) | 16 (16)
RASH (Skin and subcutaneous tissue disorders) | 47 (47) | 10 (10)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (5)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 17 (17) | 6 (6)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 19 (19) | 5 (5)
VITILIGO (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1)
FLUSHING (Vascular disorders) | 11 (11) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 7 (7) | 1 (1)
HYPOTENSION (Vascular disorders) | 20 (20) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication/presentation (manuscript, abstract or poster) to a journal/scientific meeting is sent to sponsor for review at least 1 month before submission who may delay submission by up to 90 days if it reasonably believes that publication of results may compromise its intellectual property rights or else insist that such data are removed. No single center/groups of centers may publish individually. Publication will not include confidential information without the permission of the sponsor.